CLINICAL TRIAL: NCT07209722
Title: PrEP4Her: Developing a Novel Strategy to Implement PrEP Into Women's Healthcare
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J Mugavero, MD, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008345; 5R34MH128002 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: PrEP Precriptions for Reproductive Aged Women
MeSH Terms: interventions — Pre-Exposure Prophylaxis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sexual Health-PRO: Patients seen during routine GYN clinic visit.
  Interventions: Behavioral: PrEP acronym (pre-exposure prophylaxis)
- Post visit (fidelity) survey: Patients who completed the survey outside of clinic visit
  Interventions: Behavioral: PrEP acronym (pre-exposure prophylaxis)

INTERVENTIONS:
Behavioral: PrEP acronym (pre-exposure prophylaxis) — Tracked PrEP prescriptions over 8 months among patients who completed the survey

SUMMARY:
The purpose of the study is to learn more about health care providers' experiences and perspectives on prescribing HIV pre-exposure prophylaxis, also known as PrEP. Providers and patients in gynecology clinics were interviewed and completed surveys to measure the feasibility and preference of prescribing PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Patient of UAB GYN clinic

Exclusion Criteria:

* Not a patient of UAB GYN clinic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive aged women, 18-45, who attended their regular GYN clinic visit
Sampling Method: Non-Probability Sample
Enrollment: 1377 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mugavero, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sexual Health-PRO | Post Visit (Fidelity) Survey
Started | 1135 | 242
Completed | 1135 | 242
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sexual Health-PRO | Post Visit (Fidelity) Survey | Total
Number analyzed (Participants) | 1135 | 242 | 1377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1135 | 242 | 1377
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: year] | 35 (11.5) | 35 (11.5) | 35 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1135 | 242 | 1377
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 727 | 100 | 827
  White | 235 | 140 | 375
  Hispanic | 143 | 2 | 145
  Asian | 30 | 0 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1135 | 242 | 1377

OUTCOME MEASURES:

1. Primary Outcome: PrEP Prescriptions
Description: Number of participants receiving a new PrEP prescription during the recruitment period
Time Frame: 8 months
Population: All women who received care at the GYN clinic during the study period received the PrEP4Her intervention as a component of their routine standard of gynecologic care.
Measure: Count of Participants; unit: Participants
Arm/Group | Sexual Health-PRO | Post Visit (Fidelity) Survey
Number analyzed (Participants) | 1135 | 242
Participants | 11 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Sexual Health-PRO | Post Visit (Fidelity) Survey
All-Cause Mortality (participants affected / at risk) | 0/1135 | 0/242
Serious Adverse Events (participants affected / at risk) | 0/1135 | 0/242
Other Adverse Events (participants affected / at risk) | 0/1135 | 0/242

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT07209722/Prot_SAP_000.pdf